CLINICAL TRIAL: NCT03183609
Title: Confirmatory Double-Blind Placebo-Controlled Efficacy Trial of a Gluten-Free Diet in a Subgroup of Persons With Schizophrenia Who Have High Levels of IgG Anti-Gliadin Antibodies (AGA IG)
Brief Title: Confirmatory Efficacy Trial of a Gluten-Free Diet in a Subgroup of Persons With Schizophrenia Who Have High Levels of IgG Anti-Gliadin Antibodies (AGA IG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Deanna Kelly, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00075175
Record Dates: First submitted 2017-06-07; First posted 2017-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Schizophrenia; Gluten Sensitivity; Schizo Affective Disorder
MeSH Terms: conditions — Schizophrenia; Celiac Disease; Psychotic Disorders | interventions — Flour

STUDY DESIGN:
Intervention Model Description: Randomized double blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluten (Active Comparator): 30 grams of gluten flour daily in protein shake
  Interventions: Other: Gluten Flour in Protein Shake
- Placebo (Placebo Comparator): 30 grams of rice flour daily in protein shake
  Interventions: Other: Rice Flour in Protein Shake

INTERVENTIONS:
Other: Gluten Flour in Protein Shake — 15 Grams Gluten Flour BID
  Arms: Gluten
Other: Rice Flour in Protein Shake — 15 Grams Rice Flour BID
  Arms: Placebo

SUMMARY:
This study purpose is to conduct a confirmatory double-blind randomized controlled trial in an inpatient setting of the effects of a tightly controlled gluten-free diet (GFD) to improve negative symptoms in people with schizophrenia or schizoaffective disorder who have antibodies to gliadin (AGA IgG). As part of the project investigators will also confirm outcomes such as cognitive symptoms, changes in peripheral and central inflammation as well as gut/blood brain barrier permeability.

DETAILED DESCRIPTION:
This study is a randomized double blind clinical trial being funded by NIMH. Investigators will need to enroll 40 cases with AGA IgG positivity in order to present a powered and convincing result about the efficacy of gluten withdrawal in the subpopulation of persons with schizophrenia with elevated AGA IgG levels. Investigators will recruit a minimum 50 to ensure they are well powered without question, and to account for dropouts. Investigators will use a battery of measures of peripheral and central inflammation as well as gut permeability at baseline and endpoint to confirm the relationship of these outcomes to changes in AGA IgG and symptom changes in the clinical trial. Investigators will test negative symptoms as a primary outcome but will test changes in other symptom domains such as positive symptoms. After the completion of the 5 week confirmatory study, investigators will discharge participants and follow them for 8 weeks in their own environment to test the maintenance of the effect following the stringent GFD, and provide education on gluten free shopping, cooking and eating.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV/DSM 5 diagnosis of schizophrenia or schizoaffective disorder
2. Positive for antibodies to gliadin (IgG > 20 U)
3. SANS total score ≥ 20 and the affective flattening or alogia global item ≥ 3
4. Age 18- 64 years
5. Same antipsychotic for at least 4 weeks
6. Ability to consent determined by a score of 10 or greater on the Evaluation to Sign Consent.

Exclusion Criteria:

1. Persons already on gluten free diets
2. Positivity to tissue transglutaminase (tTg) antibodies or known history of Celiac Disease
3. Pregnant or lactating females
4. Medical condition whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol
5. Meets DSM-5 criteria for alcohol or substance use disorder (other than nicotine) within the last month
6. Gluten ataxia, as measured by the Brief Ataxia Rating Scale

   Additional exclusion for those participating in optional imaging component:
7. Non-removable ferromagnetic metal on or within the body
8. Current claustrophobia
9. Inability to lie supine for 1.5 hours

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Negative symptom change as defined by difference in Clinical Assessment of Negative Symptoms -Motivation and Pleasure scale (CAINS-MAP) | 5 weeks
  This will be measured by the difference in Clinical Assessment of Negative Symptoms -Motivation and Pleasure scale CAINS-MAP) score from baseline to week 5, with a lower score yielding a better outcome.

SECONDARY OUTCOMES:
Change in cognitive function as measured by change in MATRICS Consensus Cognitive Battery (MCCB) | 5 weeks
  This will be measured by the difference in MATRICS Consensus Cognitive Battery (MCCB) scores from baseline to week 5

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Psychiatric Research Center (MPRC) Outpatient Research Program (ORP); the MPRC Treatment Research Program (TRP), Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daniels EC, Eaton WW, Cihakova D, Talor MV, Lemke H, Mo C, Chen S, Notarangelo FM, Rodriguez KM, Kelly DL. The relationship of peripheral inflammation with antibodies to gliadin (AGA IgG) in persons with schizophrenia. Schizophr Res. 2023 Jun;256:50-51. doi: 10.1016/j.schres.2023.02.027. Epub 2023 May 5. No abstract available. PMID 37150147
- See also: Maryland Psychiatric Research Center — http://www.mprc.umaryland.edu